CLINICAL TRIAL: NCT04209504
Title: Evaluating Hemidiaphragmatic Paralysis With Prolonged Neural Blockade From an Interscalene Brachial Plexus Block
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104053
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Surgery; Shoulder Pain; Shoulder Injuries; Shoulder Arthritis; Shoulder Disease; Rotator Cuff Tears; Rotator Cuff Injuries; Rotator Cuff Arthropathy of Left Shoulder; Rotator Cuff Arthropathy of Right Shoulder; Rotator Cuff Repair
Keywords: Rotator Cuff Repair; Shoulder Surgery; Hemidiaphragmatic paralysis; Interscalene Block; Interscalene Catheter; Interscalene Liposomal Bupivacaine
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries; Rotator Cuff Injuries | interventions — Ultrasonography; Ropivacaine; Bupivacaine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Continuous Perineural Catheter: Placement of preoperative continuous perineural catheter using 25 milliliters (mL) 0.5% ropivacaine with 1:400,000k ropivacaine for initial block and 0.2% ropivacaine for continuous infusion.
  Interventions: Diagnostic Test: Ultrasound; Drug: Ropivacaine; Device: MediPines AGM100 Advanced Respiratory Monitoring System
- 10 mL Liposomal Bupivacaine Single Shot: Placement of preoperative single shot using 10mL liposomal bupivacaine (Exparel; n=20) plus 5 mL 0.5% bupivacaine
  Interventions: Diagnostic Test: Ultrasound; Drug: Bupivacaine; Device: MediPines AGM100 Advanced Respiratory Monitoring System
- 20 mL Liposomal Bupivacaine Single Shot: Placement of preoperative single shot using 20mL liposomal bupivacaine (Exparel; n=20) plus 5 mL 0.5% bupivacaine
  Interventions: Diagnostic Test: Ultrasound; Drug: Bupivacaine; Device: MediPines AGM100 Advanced Respiratory Monitoring System

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound guided evaluation of diaphragm ipsilateral to the block side.
Drug: Ropivacaine — Local anesthetic (numbing drug)
  Other Names: Naropin
  Groups: Continuous Perineural Catheter
Drug: Bupivacaine — Local anesthetic (numbing drug)
  Other Names: Liposomal bupivacaine; Exparel; Marcaine
  Groups: 10 mL Liposomal Bupivacaine Single Shot; 20 mL Liposomal Bupivacaine Single Shot
Device: MediPines AGM100 Advanced Respiratory Monitoring System — Non-invasive respiratory monitor to measure oxygenation and ventilation parameters
  Other Names: non-invasive respiratory monitor

SUMMARY:
This prospective observational study aims to evaluate the incidence of hemidiaphragmatic paralysis in patients receiving interscalene brachial plexus nerve block with prolonged neural blockade. English speaking American Society of Anesthesiologists (ASA) 1-3 patients ages 18-80 receiving prolonged interscalene nerve block will be randomized into 3 groups: first group receiving a perineural catheter infusing 0.2% ropivacaine; the second group receiving a single shot injection of 10mL liposomal bupivacaine (Exparel; n=20) plus 5 mL 0.5% bupivacaine and the third receiving 20mL liposomal bupivacaine plus 5mL bupivacaine (to be determined by the attending anesthesiologist).Primary outcome will be incidence of hemidiaphragmatic paralysis postoperative day 1 as measured by point of care (POCUS) ultrasound.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate the incidence of hemidiaphragmatic paralysis in patients receiving interscalene brachial plexus nerve block with prolonged neural blockade. English speaking ASA 1-3 patients ages 18-80 receiving prolonged interscalene nerve block will be randomized into 3 groups first group receiving a perineural catheter infusing 0.2% ropivacaine; the second group receiving a single shot injection of 10mL liposomal bupivacaine (Exparel; n=20) plus 5 mL 0.5% bupivacaine and the third group receiving 20mL liposomal bupivacaine plus 5mL bupivacaine (to be determined by the attending anesthesiologist). Primary outcome will be incidence of hemidiaphragmatic paralysis postoperative day 1 as measured by point of care (POCUS) ultrasound. Secondary outcomes include incidence of hemidiaphragmatic paralysis as measured by point of care ultrasound (POCUS) in the immediate postoperative period, postoperative day (POD) 1, POD2, and POD3 and noninvasive measures of pulmonary gas exchange at pre-op, post-op, POD1, POD2, and POD3. Additionally, the investigators will look at pain scores (scale of 0-10) and opioid consumption (in oral morphine equivalents) at previously defined time points listed above. Furthermore, the investigators will record known side effects of interscalene blocks including hoarseness and Horner's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* English speaking 18-80 year old ASA 1-3 patients
* Primary shoulder surgery
* Must live within a 25 mile radius

Exclusion Criteria:

* ASA 4 or 5
* Revision shoulder surgery
* Diagnosis of chronic pain
* Daily chronic opioid use (over 3 months of continuous opioid use)
* Inability to communicate pain scores or need for analgesia
* Infection at the site of block placement
* Age under 18 years old or greater than 80 years old
* Pregnant women (as determined by point-of-care serum bHCG)
* Intolerance/allergy to local anesthetics
* Weight <50 kg
* BMI > 40
* severe pulmonary disease including chronic obstructive pulmonary disease and restrictive lung disease
* Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance.
* Current or historical evidence of any clinically significant disease or condition that, in the opinion of the investigator, may increase the risk of surgery or complicate the subject's postoperative course.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ages 18-80 undergoing shoulder surgery per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Hemidiaphragmatic paralysis - ipsilateral - postoperative day (POD) 1 | 24 hours
  Ultrasound guided evaluation of ipsilateral hemidiaphragmatic paralysis POD1

SECONDARY OUTCOMES:
Hemidiaphragmatic paralysis - ipsilateral - PACU, POD2, POD3 | up to 72 hours
  Ultrasound guided evaluation of ipsilateral hemidiaphragmatic paralysis in PACU, POD2, and POD 3
Noninvasive pulmonary measures of gas exchange | up to 72 hours
  Noninvasive pulmonary measures of gas exchange
Pain scores | up to 72 hours
  Numerical Rating Scale (NRS) 11 pain scores (0-10; 0=no pain, 10=worst pain ever) at Post Anesthesia Care Unit (PACU), POD1, POD2, POD3
Opioid consumption | up to 72 hours
  Opioid consumption in Oral Morphine Equivalents (OMEs) at PACU, POD1, POD2, POD3
Hoarseness | up to 72 hours
  Incidence of recurrent laryngeal nerve palsy (subjective)
Horner's Syndrome | up to 72 hours
  Incidence of Horner's Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Kumar, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared; patients will be deidentified and no personal information or medical records used once patient has completed the study.